CLINICAL TRIAL: NCT03272815
Title: Evaluation of a Novel Point-of-care Percussion Device (PD) for Detection of Pneumothorax in Patients Following Thoracic Surgery
Brief Title: Percussion Device (PD) for Detection of Pneumothorax
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device requires further modification
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard Malthaner, Thoracic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 109205
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Pneumothorax
Keywords: pneumothorax; chest tube removal; percussion
MeSH Terms: conditions — Pneumothorax | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: A prospective clinical feasibility cohort study.
Who Masked: Outcomes Assessor
Masking Description: Radiologists are unaware of the intervention or the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD arm (Experimental): Patients undergoing assessment of the chest with the percussion device (PD).
  Interventions: Device: Percussion Device (PD)
- US arm (Active Comparator): Patients undergoing assessment of the chest with the ultrasound (US).
  Interventions: Device: Ultrasound (US)

INTERVENTIONS:
Device: Percussion Device (PD) — A laboratory prototype of the Percussion Device (PD) has been designed and built; laboratory data collection software, signal analysis and classification algorithms have been developed. It has been designed to detect a pneumothorax.
  Arms: PD arm
Device: Ultrasound (US) — The SonoSite hand help portable ultrasound device.
  Arms: US arm

SUMMARY:
This study aims to examine the safety and efficacy of the Percussion Device in detecting a pneumothorax in patients that have undergone thoracic surgery.

DETAILED DESCRIPTION:
A prospective, non-randomized clinical feasibility cohort study. The purpose of this feasibility study is to collect preliminary performance and safety information for the Percussion Device (PD). Patients satisfying the inclusion criteria will be approached for study enrolment before their surgery in clinic. Following surgery and after the patient's chest tube has been removed, evaluation of the chest using the PD and ultrasound will be performed by two independent assessors (a nurse practitioner or resident on the Thoracic Surgery Team) prior to the post-removal CXR. Details of study procedure are details in section 2.8. The PD's performance metric will be compared against CXR results, which is considered the gold standard in diagnosing a pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* All patients that have undergone an open or thoracoscopic thoracic procedure requiring a chest tube at London Health Sciences Centre (LHSC), London, Ontario.

Exclusion Criteria:

* Patients less than 18 years old Patients unable to consent Patients with known persistent pneumothorax prior to chest tube removal Patients who are pregnant Patients with severe chest wall deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Performance metrics | 2 years
  Performance metrics of the PD in detecting the presence of a pneumothorax following the removal of the last chest tube in patients that have undergone thoracic surgery compared to the CXR reported by a blinded radiologist unaware of the study.

SECONDARY OUTCOMES:
Inter-rater reliability | 2 years
  The secondary outcomes will include inter-rater reliability with the PD or ultrasound or CXR.
Adverse Events | 2 years
  Any adverse event associated with the PD or ultrasound or CXR.
Marginal Costs | 2 years
  Marginal costs differences between the surgeon performed PD and CXR will be based on an overall risk-benefit assessment that will take into account accuracy and costs of facilities as well as physician services.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Malthaner, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No